CLINICAL TRIAL: NCT06286436
Title: Effect of Dual-task Training on the Number of EEG Band in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Mahia Physiotherapy Clinic (Qom, Iran) (Unknown)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, Head of iHealthy Research Group, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR.SBMU.RETECH.REC.1401.842
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Electroencephalography
Keywords: Electroencephalography; rehabilitation; physiotherapy; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual-task training (Experimental)
  Interventions: Other: Dual-task training

INTERVENTIONS:
Other: Dual-task training — The intervention will consist of three different tasks that participants have to carry out while performing mental calculations (counting backwards from 100 by ones, twos, and threes). The three tasks will be as follows: grouping blocks of different colours into groups according to colour; picking up beans with a spoon and carrying them to a specific place; opening and closing a bottle cap with the affected hand. The total duration of the intervention will be 12 sessions, divided into three days per week for four weeks.

SUMMARY:
Stroke is a prevalent global health concern, causing widespread disability as it disrupts blood supply to the brain, leading to functional impairments. Upper limb dysfunction affects over 80% of stroke survivors acutely and becomes permanent in approximately 60%, hindering daily activities and autonomy. Dual-task training (DTT), involving simultaneous cognitive and motor tasks resembling daily activities, is proposed as an effective intervention.

The study suggests using electroencephalogram (EEG) analysis, particularly the Fast Fourier Transform (FFT), to assess changes in brain signals pre- and post-DTT intervention. EEG provides real-time insights into brain function, and FFT analyzes signal frequencies. The intervention involves three tasks performed concurrently with mental calculations, such as sorting blocks and manipulating objects. This 12-session, four-week intervention aims to improve upper limb function. The study explores EEG's role in evaluating DTT effects on stroke patients, particularly using FFT to analyze brain signal frequencies.

DETAILED DESCRIPTION:
Stroke is one of the most common diseases and causes of disability worldwide. This condition occurs when the blood supply to the brain tissue is disrupted, leading to ischaemia of the brain tissue and the functional impairments in the different systems of the body that this entails. One of the most prevalent and disabling dysfunctions in stroke patients is that related to the upper limb, with more than 80% experiencing this condition acutely and being permanent in approximately 60% of stroke survivors despite rehabilitation. The alteration of the functionality of the upper limbs of the person after stroke, including muscle weakness, sensory disorders, increased muscle tone and lack of neuromuscular control and coordination means that the person is not able to carry out normal activities of daily living (ADLs), thus affecting their autonomy and independence.

Most ADLs often require a combination of cognitive and motor tasks at the same time. These tasks are especially difficult for people who have suffered a stroke as their mental and physical capacity is impaired and therefore performing more than one task becomes a challenge. On the other hand, dual-task training (DTT) understood as a treatment method based on exercises involving 2 or more tasks at the same time related to the person's ADLs can be a interesting approach to improve the above mentioned upper limb disorders.

One of the tools recommended to analyse how a treatment or intervention affects the central nervous system of the person with stroke is the electroencephalogram (EEG), as it provides a continuous, real-time, non-invasive measurement of brain function that provides new insights into the pathophysiology of the brain. EEG analysis of brain disorders can be carried out with different methods such as network analysis and connectivity examination, machine learning, graph neural networks and examination of band frequency changes.

Among the EEG analysis methods that have not yet been tested in the stroke population following DTT intervention is the Fast Fourier Transform (FFT), a powerful tool for analysing the frequency of signals. When applied to a signal, the FFT function converts the signal from a time domain to a frequency domain. The main objective of this study is to analyse how in the different EEG bands (delta, theta, alpha and beta) of stroke patients are modified after converting the brain signal into Fourier series/transforms before and after a DTT intervention.

The intervention will consist of three different tasks that participants have to carry out while performing mental calculations (counting backwards from 100 by ones, twos, and threes). The three tasks will be as follows: grouping blocks of different colours into groups according to colour; picking up beans with a spoon and carrying them to a specific place; opening and closing a bottle cap with the affected hand. The total duration of the intervention will be 12 sessions, divided into three days per week for four weeks.

The main outcome is EEG data, which will be collected both before and after intervention, under the supervision of a neurologist, with the participant in a resting state and eyes closed. EEG recording is carried out during 3 minutes with 10-20 system, 19 electrodes (Fp1, Fp2, F7, F3, Fz, F4, F8, T7, C3, Cz, C4, T8, T10, P3, Pz, P4, P8, T9, P7) and a sampling rate of 256 Hz. The Fast Fourier Transform (FFT), which has proven to have less order complexity, will be used for the data analysis.

In addition, other variables on upper limb function, elbow flexor muscle tone, wrist extension range of motion and handling in activities of daily living will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke proven by imaging evidence
* Women between 35 and 75 years old
* At least six months have passed since the onset of the stroke

Exclusion Criteria:

* Suffering from another neurological or orthopedic disease
* Score greater than 3 on the modified modified Ashworth scale in the upper limb
* Having received a botulinum toxin injection before or during the course of the study
* History of brain surgery
* Be using medication that may alter cortical activity or brain plasticity or aimed at reducing the level of spasticity.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
EEG Data | Before and after intervention (4 weeks)
  EEG data will be collected both before and after intervention, under the supervision of a neurologist, with the participant in a resting state and eyes closed. EEG recording will be carried out during 3 minutes with 10-20 system, 19 electrodes (Fp1, Fp2, F7, F3, Fz, F4, F8, T7, C3, Cz, C4, T8, T10, P3, Pz, P4, P8, T9, P7) and a sampling rate of 256 Hz. Frequencies below 1Hz and above 40Hz will be filtered. One of the three minutes of EEG collection will be randomly selected, and analysis will be carried out for that minute only. Before data analysis, abnormal waves such as blinking and electromyographic signals will be removed. All these operations will be carried out in MATLAB and by EEGLab toolbox.

SECONDARY OUTCOMES:
Upper limb function | Before and after intervention (4 weeks)
  Upper limb function will be measure with the "Box and Block test", which is a functional test to specifically measure unilateral manual dexterity including grasping, carrying and releasing objects, consisting of transferring 150 coloured wooden cubes, each measuring 1 inch, from one box to another as quickly as possible within 60 seconds using only the affected hand.
Elbow flexor muscle tone | Before and after intervention (4 weeks)
  Elbow flexor muscle tone will be measured with the modified modified Ashworth scale, scored on an ordinal scale from 0 to 4: 0 = no increase in muscle tone; 1 = slight increase in muscle tone, manifested by a catch and release or minimal resistance at the end of the range of motion when affected part is moved in flexion or extension; 2 = a marked increase in muscle tone, manifested by a catch in the middle range and resistance throughout the remainder of the range of motion, but the affected part easily moved; 3 = considerable increase in muscle tone, passive movement difficult; and 4 = affected part rigid in flexion or extension
Wrist extension range of motion | Before and after intervention (4 weeks)
  Wrist extension range of motion will be measured with a goniometer
ADLs | Before and after intervention (4 weeks)
  The functional assesment of the patient in ADLs will be measured with the Barthel Index, which is a scale that scores ten basic aspects of activity related to self-care and mobility (bowels, bladder, grooming, toilet use, feeding, transfer, mobility, dressing, stairs and bathing) from 0 to 100 where lower scores indicate greater dependency

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Beheshti University of Medical Sciences, Tehran, Velenjak, Iran

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once research has been published